CLINICAL TRIAL: NCT01468064
Title: Autologous Bone Marrow Stromal Cell and Endothelial Progenitor Cell Transplantation in Patients With Ischemic Stroke: a Randomized Controlled Trial
Brief Title: Autologous Bone Marrow Stromal Cell and Endothelial Progenitor Cell Transplantation in Ischemic Stroke
Acronym: AMETIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Collaborators: The Second People's Hospital of Nanhai District of Foshan (Unknown); The First People's Hospital of Haizhu District Guangzhou (Other); Cellonis Biotechnology Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Zhen-Zhou Chen, Department of Neurosurgery, Zhujiang Hospital, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZJH-001; 2011A030400007 (Other Grant/Funding Number: The Key project of Guangdong Science and Technology Program)
Record Dates: First submitted 2011-11-02; First posted 2011-11-09 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Stroke; Infarction, Middle Cerebral Artery
Keywords: Central Nervous System Diseases; Stroke; Infarction, Middle Cerebral Artery; Cerebral Infarction; Cerebrovascular Accident; Stem Cell Transplantation; Mesenchymal Stem Cell Transplantation; Bone marrow stromal cells; Mesenchymal Stem Cells; Endothelial progenitor cells; Adult Stem Cells; Cell Therapy
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery; Central Nervous System Diseases; Cerebral Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BMSCs group (Experimental)
  Interventions: Genetic: Autologous BMSCs transplantation
- EPCs group (Experimental)
  Interventions: Genetic: Autologous EPCs transplantation
- Control group (Placebo Comparator)
  Interventions: Genetic: IV infusion of placebo

INTERVENTIONS:
Genetic: Autologous BMSCs transplantation — The first transplantation: 2.5 million cells per kg autologous BMSCs suspended in 100 ml saline plus 5% autologous serum are infused intravenously approximately 4 weeks after bone marrow aspiration.
  The second transplantation: the same amount of cells are again transplanted approximately 1 weeks after initial boosting.
  Other Names: Autologous Bone marrow stromal cells transplantation; Autologous Mesenchymal stem cells transplantation
  Arms: BMSCs group
Genetic: Autologous EPCs transplantation — The first transplantation: 2.5 million cells per kg autologous EPCs suspended in 100 ml saline plus 5% autologous serum are infused intravenously approximately 4 weeks after bone marrow aspiration.
  The second transplantation: the same amount of cells are again transplanted approximately 1 weeks after initial boosting.
  Other Names: Autologous endothelial progenitor cells transplantation
  Arms: EPCs group
Genetic: IV infusion of placebo — IV infusion of saline plus 5% autologous serum.
  Other Names: Placebo control group
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the feasibility, efficacy, and safety of autologous transplantation of ex vivo expanded bone marrow stromal cells (BMSCs)and endothelial progenitor cells (EPCs) for treatment of patients with ischemic stroke.

DETAILED DESCRIPTION:
This study is a multi-center, single-blind, randomized, parallel controlled trail. Patients with acute cerebral infarcts within the middle cerebral arterial territory and with severe neurological deficits will be enrolled and randomly allocated into 3 groups: autologous BMSCs transplantation group, autologous EPCs transplantation group and Placebo control group. Randomization codes were established by the study statistician and were revealed only to the stem cell laboratory technician responsible for separating the cells into aliquots or preparing the placebo material. All patients will undergo a Bone Marrow aspiration procedure at 7 days after symptom onset. BMSCs and EPCs will be expanded ex vivo and then intravenously infused into own body, respectively. The control group will not receive cell therapy. Observe will followed for up to 1 year after the onset. Neurological score, neuroimaging, mortality of any cause, side effects, and new-onset comorbidities will be monitored and compared between each groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years, within 7 days of the onset of symptoms
2. Ischemic lesion within the MCA territory as assessed using diffusion-weighted imaging (DWI)
3. The National Institutes of Health Stroke Scale (NIHSS) ≥ 7 at day 7 after the onset
4. Signed informed consent

Exclusion Criteria:

1. Lacunar syndrome
2. Diagnosis other than ischemic stroke(eg. Intracranial hemorrhage or Intracranial tumor)
3. Hematological causes of stroke
4. Severe respiratory, hepatic, or renal disorders
5. Presence of severe febrile illness or viral diseases
6. Malignant diseases
7. Presence of autoimmune diseases
8. Positive response of penicillin skin test, or multiple drug allergies
9. Breast-feeding or pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of adverse events after infusion of BMSCs or EPCs. | 1 year

SECONDARY OUTCOMES:
Changes in functional outcomes measured by the modified Rankin Scale (mRS) and the Barthel index (BI). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhou Chen, MD., phD., Principal Investigator — Department of Neurosurgery, Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lee JS, Hong JM, Moon GJ, Lee PH, Ahn YH, Bang OY; STARTING collaborators. A long-term follow-up study of intravenous autologous mesenchymal stem cell transplantation in patients with ischemic stroke. Stem Cells. 2010 Jun;28(6):1099-106. doi: 10.1002/stem.430. PMID 20506226
- [Background] Bang OY, Lee JS, Lee PH, Lee G. Autologous mesenchymal stem cell transplantation in stroke patients. Ann Neurol. 2005 Jun;57(6):874-82. doi: 10.1002/ana.20501. PMID 15929052
- [Derived] Fang J, Guo Y, Tan S, Li Z, Xie H, Chen P, Wang K, He Z, He P, Ke Y, Jiang X, Chen Z. Autologous Endothelial Progenitor Cells Transplantation for Acute Ischemic Stroke: A 4-Year Follow-Up Study. Stem Cells Transl Med. 2019 Jan;8(1):14-21. doi: 10.1002/sctm.18-0012. Epub 2018 Aug 29. PMID 30156755